CLINICAL TRIAL: NCT01606020
Title: Effects of Sleep Deprivation on Driving Performance and Central Fatigue
Brief Title: Sleep Deprivation : Effects on Driving Performance and Central Fatigue
Acronym: PrivSom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1108128; 2011-A00895-36 (Other: AFSSAPS)
Record Dates: First submitted 2012-05-03; First posted 2012-05-25 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Healthy Volunteers
Keywords: effects of sleep deprivation; Transcranial Magnetic Stimulation; male, healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep deprivation First (Active Comparator): First night D7 :
  Overnight, the subjects stay in their homes (reading, watching TV, playing cards). Two experimenters will take turns to never leave them alone and avoid any micro-sleep.
  Second night D28 :
  Overnight, the subjects stay in their homes. No intervention during this night.
  Interventions: Other: sleep deprivation; Other: No intervention
- sleep deprivation second (Active Comparator): First night D7 :
  Overnight, the subjects stay in their homes. No intervention during this night.
  Second night D28 :
  Overnight, the subjects stay in their homes (reading, watching TV, playing cards). Two experimenters will take turns to never leave them alone and avoid any micro-sleep.
  Interventions: Other: sleep deprivation; Other: No intervention

INTERVENTIONS:
Other: sleep deprivation — Overnight, the subjects stay in their homes (reading, watching TV, playing cards). Two experimenters will take turns to never leave them alone and avoid any micro-sleep.
Other: No intervention — Overnight, the subjects stay in their homes. No intervention during this night

SUMMARY:
The effects of sleep deprivation (SD) on performance, while contradictory at first glance, are in reality rather clear when exercise duration is considered, i.e. intense/supramaximal versus prolonged exercises. This latter type of exercise leads to the most important performance decrements after SD.

DETAILED DESCRIPTION:
The effects of sleep deprivation (SD) on performance, while contradictory at first glance, are in reality rather clear when exercise duration is considered, i.e. intense/supramaximal vs. prolonged exercises. This latter type of exercise leads to the most important performance decrements after SD. However, the causes of this accentuated fatigability in endurance exercise with sleep deficit are not known. Several hypotheses have been proposed such as lower pH before exercise, lower ventilation due to depreciated response to hypercapnia/hypoxia, or haemodilution. Yet the most plausible explanation is a lower tolerance to prolonged exercise because SD increases the rate of perceived exertion. Another potential effect of SD is an alteration of central command during exercise. The literature is rather scarce on this topic and is only based on a few animal studies. In humans, no effect of SD on maximal strength has been reported so that maximal voluntary activation should in theory not be altered. Transcranial Magnetic Stimulation (TMS), that allows to induce a motor response from its cortical origin (and to measure the resulting contraction), is a promising tool to explore neuromuscular function. TMS has been used only in three studies after SD, none of them involving exercise and none of them measuring mechanical responses (i.e. only EMG responses, such as motor evoked potential, were measured). In addition, the results of these three studies are contradictory. The effects of SD on central fatigue (i.e. increase of the activation deficit during exercise) have never been investigated. The goal of this experiment is thus to test the hypothesis that an increase in central fatigue (at supraspinal level) in SD can participate to performance alteration during a prolonged exercise. For that purpose, measurements of neuromuscular function particularly dedicated to assess central fatigue will be performed before and after SD but also when combining SD and a fatiguing exercise conducted until exhaustion.

ELIGIBILITY:
Inclusion Criteria:

* no smoking and drugs
* regular physical activity

Exclusion Criteria:

* insufficiency cardiac or respiratory
* carrying a cardiac pacemaker

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
change value of the level of maximal voluntary activation of quadriceps muscle supraspinal | at Day 7 and Day 28
  change value of the level of maximal voluntary activation of quadriceps muscle supraspinal between before and after endurance exercise after a night of sleep deprivation

SECONDARY OUTCOMES:
variation of the activation level of excitability and supraspinal / cortical | At Day 7 and Day 28
  variation of the activation level of excitability and supraspinal / cortical inhibition after a night of sleep deprivation
level variation in test performance from test of Simon | At Day 7 and Day 28
  level variation in test performance from test of Simon before, during and after endurance exercise following a night of sleep deprivation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MILLET, PhD, Study Chair — Jean Monnet University
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France